CLINICAL TRIAL: NCT04145882
Title: Is it Better to Add Supination Osteotomy, Varisation Osteotomy, or Both to Distal Chevron as Part of Hallux Valgus Management : a Prospective Randomized Trial
Brief Title: Efficacy of Additional Osteotomies to Correct Hallux Valgus
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Elsan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CPL-2019-HV
Record Dates: First submitted 2019-10-29; First posted 2019-10-31 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Hallux Valgus
MeSH Terms: conditions — Hallux Valgus

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- No additional osteotomy (Active Comparator)
  Interventions: Procedure: additional osteotomies
- varisation osteotomy addition (Experimental)
  Interventions: Procedure: additional osteotomies
- supination osteotomy addition (Experimental)
  Interventions: Procedure: additional osteotomies
- both (varisation + supination) osteotomies addition. (Experimental)
  Interventions: Procedure: additional osteotomies

INTERVENTIONS:
Procedure: additional osteotomies — varisation osteotomy, supination osteotomy or both

SUMMARY:
Deviation of the big toe in valgus at the level of the first metatarsophalangeal joint is called Hallux Valgus. In case of significant pain especially due to a conflict with the shoes, surgery could be indicated. Angle between the first metatarsal (M1) and the first phalangeal (P1) is named Hallux Valgus Angle (HVA). Angle between M1 and the second metatarsal (M2) is named InterMetatarsal Angle (IMA). Angle between M1 distal articular surface and M1 shaft axis in a frontal plane is named Distal Metatarsal Articular Angle (DMAA).

Insufficient surgical correction is a risk factor of recurrence (HVA>20° after surgery). According to Okuda et al in a 67 patients group treated by proximal osteotomies correction, postoperative risk factors of recurrence at 33 month of follow-up are : HVA>40° before the surgery and HVA>15° with an IMA>10° 10 weeks (3-24) after the surgery.

Currently, one of the most common used procedure is a translated (laterally) distal chevron associated with a release of the metatarso-sesamoid suspensory ligament and a Akin procedure on P1. Nevertheless this procedure does not correct deformation in all plans. HVA and IMA are corrected but DMAA and M1 pronation angle are not.

Surgeons can add three different osteotomies in this type of chevron. In the dorsal saw cut a varisation wedge osteotomy is possible , in the plantar saw cut a supination wedge osteotomy is possible, and both are possible. No studies have tried to assess these three possibilities.

The investigators hypothesize that the addition of a varisation and/or a supination wedge osteotomies in a distal chevron decrease risk factors of recurrence at six months of follow-up

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 18 years.
* Informed consent

Exclusion Criteria:

* Associated lesser metatarsals surgery.
* Associated surgery on midfoot, hindfoot or ankle.
* Neurologic diseases (Charcot Marie Tooth disease, poliomyelitis, compartment syndrome sequelae)
* Clinical or X-ray degenerative signs (Hallux rigidus) or irreducible deformations (MTP1 arthrodesis indications).
* Patient who declined the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 515 (Actual)
Dates: Start 2019-09-11 (Actual); Primary Completion 2021-07-29 (Actual); Study Completion 2026-09-11 (Estimated)

PRIMARY OUTCOMES:
Rate of patients having both Hallux Valgus Angle >15° and InterMetatarsal Angle >10° | 6 months
  on weight bearing X-Rays

SECONDARY OUTCOMES:
Recurrence of hallux valgus (HVA>20°). | 5 years
American Orthopedic Foot and Ankle Forefoot Score (AOFAS) | 6 months
  Mini 0 (Worse) - Maxi 100 (Better)
American Orthopedic Foot and Ankle Forefoot Score (AOFAS) | 5 years
  Mini 0 (Worse) - Maxi 100 (Better)
Patient satisfaction (Likert scale) | 6 months
  very satisfied/satisfied/fairly satisfied/no satisfied
Patient satisfaction (Likert scale) | 5 years
  very satisfied/satisfied/fairly satisfied/no satisfied

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Clinique Lille sud, Lesquin
  - Clinique du Parc Lyon, Lyon
  - Clinique Mégival, Saint-Aubin-sur-Scie
  - Clinique de l'Union, Saint-Jean

IPD SHARING:
Plan to Share IPD: No